CLINICAL TRIAL: NCT03719807
Title: A Protocol of Accelerated Rehabilitation for Patients Undergoing Adolescent Idiopathic Scoliosis Correction Surgery - An Internal Pilot Study
Brief Title: Protocol of Accelerated Rehabilitation Following Surgical Correction of Adolescent Idiopathic Scoliosis
Acronym: PARIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ROH18ORTH07
Record Dates: First submitted 2018-10-11; First posted 2018-10-25 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2018-10

CONDITIONS: Scoliosis Idiopathic
Keywords: rehabilitation; post-operative; scoliosis correction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Usual Care No routine outpatient physiotherapy following discharge home post-operatively in line with standard care.
  Interventions: Other: Usual Care
- Intervention Group (Experimental): 12 x Exercise//Rehabilitation sessions Begin at 6 weeks. 6 x weekly sessions Followed by 6 x bi-weekly sessions In line with Accelerated Rehabilitation protocol
  Interventions: Other: Rehabilitation protocol

INTERVENTIONS:
Other: Rehabilitation protocol — A physiotherapy rehabilitation protocol - comprising of pragmatic exercises.
  Arms: Intervention Group
Other: Usual Care — No routine outpatient physiotherapy. Normal inpatient physiotherapy to match intervention group.
  Arms: Control Group

SUMMARY:
This study aims to identify whether an accelerated physiotherapy led rehabilitation programme for adolescents undergoing idiopathic scoliosis correction surgery can be delivered safely and effectively post-operatively, and whether it might improve activity levels and quality of life outcomes for the study group.

This research is being conducted as previous research indicates that up to 41% of patients who have surgical correction of their scoliosis either return to athletic activity at a lower level than before, or they do not return to athletic activity at all. This is despite significant advancement in the instrumentation being used in recent years which makes the corrections more stable and robust. Some studies have shown that surgically treated AIS patients have significantly reduced physical function and quality of life scores, and that this could be improved with exercise. So far no trials have investigated whether post-operative rehabilitation can improve quality of life for these patients.

The initial study will be a pilot study, comprising of 20 participants in a small, pragmatic randomised controlled trial (RCT). It will be conducted at The Royal Orthopaedic Hospital, a specialist National Health Service (NHS) orthopaedic centre. Adolescents (between 11-18 years of age) who have a diagnosis of adolescent idiopathic scoliosis (AIS) and are on the waiting list for surgical correction of this scoliosis will be included. The study will compare a post-operative accelerated rehabilitation programme (commenced at 6 weeks post surgery) with usual care and investigate if the accelerated intervention can be delivered safely and effectively after this procedure. Following surgery, both groups will have the same inpatient rehabilitation up until the point of discharge home. The intervention group will then complete 12 sessions of physiotherapy as an outpatient, which starts at 6 week post-op. The usual care group will not have any further physiotherapy, in line with current standard practice at this centre. Both groups will be assessed using patient reported outcome measures pre-operatively, and at 6 months and 12 months post-operatively, to assess function and quality of life.

DETAILED DESCRIPTION:
This is an internal pilot study, comprising a small pragmatic, RCT conducted at the Royal Orthopaedic Hospital NHS Foundation Trust. It will aim to test whether an accelerated rehabilitation protocol can be implemented safely and effectively for patients following correction surgery for AIS and, if so, whether the intervention leads to an improvement in activity levels or quality of life scores in the study group. It will also aim to identify whether it is feasible to implement such a programme as part of a bigger RCT in the future based on the attendance rate and functional improvements.

Recruitment:

Participants will be identified and recruited pre-operatively through the spinal deformity waiting list. The Eligibility of participants can be obtained through their medical notes.

Once identified and confirmed as eligible, participants will be approached by one of the research nurses and invited to take part in the study. There are two potential pathways to recruitment:

* If the participant is due to have a clinic appointment (such as a pre-operative assessment) within one month of their surgery, then patient information sheets and study invitation letters will be given to them at this appointment with their normal pre-operative information, by a research nurse. Follow up telephone calls can be conducted 7-10 days later to give participants and parents time to read and consider the information. Consent can be obtained at subsequent pre-operative appointments if any are scheduled (giving participants time to consider before consent), or at the time of admission for surgery should the participant want more time to consider.
* If the patient has already completed their pre-operative assessment and is not due to attend for any further appointments prior to their surgery, they will be sent this information in the post. Participants will be given adequate time to read and consider the information given. This time scale has been set at 7-10 days, to give participants and their parents plenty of time to read the information and consider it before contacting them. A telephone call will then take place prior to their admission to ask whether they have read and had time to consider the information and whether they have any questions. If they would like to take part in the trial, then a research clinician will meet with them the day before their surgery, when they are admitted, in order to fill in the consent form and to fill in the baseline questionnaire.

Evidence of screening for all potential participants, whether recruited or not, should be kept and recorded.

Post-Operatively:

Following their surgery, a research clinician will visit the participant on the ward, approximately 3-4 days after their surgery. This is to check from the operation records that there has not been any surgical complications that would exclude them from the study, and to check that the participant and their parents are still happy to take part in the study. If so, the participant will be randomised by the research clinician at this point. Randomisation will be performed using sealed envelopes. The results of the randomisation will be given to the treating physiotherapist. Prior to the participants discharge home from the ward, the treating physiotherapist will inform the participant which group they have been allocated to. If they are in the intervention arm their outpatient physiotherapy appointments will be booked for them at this point. If they are randomised to the usual care arm, then the patient will be discharged from the ward and will not be required to attend for any further physiotherapy. All patients will have the same level of inpatient care on the ward prior to discharge home.

Intervention:

There are two arms to the trial and there will be 10 participants randomly allocated to each arm. The control group will be seen by the physiotherapist on the ward and given daily physiotherapy up until the point of discharge home. They will then not have any further physiotherapy follow up, as part of usual care, unless there are any post-operative complications that require a physiotherapy referral. If a participant in the control group is referred back into secondary care for physiotherapy during the trial, then this will be recorded as a deviation from the protocol and included in final analysis.

The intervention group involves the same inpatient care as the control arm, plus 12 sessions of physiotherapy as an outpatient, and this will start 6 week post-operatively. The participants will initially come once a week for 6 weeks. Then from 12 weeks post-operatively they will be required to come once every 2 weeks. The treatment will be pragmatic depending on the patients individual goals and needs, but will follow the accelerated rehabilitation protocol that has been agreed with the spinal deformity consultant surgeons. Once the participants in the intervention arm have completed their 12 sessions, they will be discharged from physiotherapy for self-management, unless they have any on-going physiotherapy related needs. In this case they can continue with physiotherapy and it will be recorded as a deviation from the protocol.

Data Collection and Follow Up:

All 20 participants will fill in a baseline data collection booklet at the time of consent, which is just before their surgery. This includes patient reported outcome measures. All participants in both groups will be followed up at approximately 6 months, and again at 12 months, following their surgery. Where possible, participants will be approached at their 6 month and 12 months consultant review appointments to fill out the questionnaires for data collection. If this is not possible, then the questionnaires will be sent out in the post for them to complete and return to the research department. The questionnaires booklets contain:

Data will also be collected regarding recruitment rates, compliance with the intervention and serious adverse events (SAEs).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 11-18 years old at the time of surgery.
* Diagnosis of AIS confirmed by spinal deformity team.
* On the waiting list to have a posterior or combined anterior/posterior scoliosis correction surgery.

Exclusion Criteria:

* Underlying cause of scoliosis which makes it not idiopathic.
* Significant post-operative complications that prevents participation in the trial.
* Any significant learning disabilities or cognitive impairment that would limit the patient's ability to take part in the rehabilitation protocol.
* Planned anterior-only scoliosis correction surgery.
* Patients that are unable to understand verbal instructions or written information given in English.
* Patients involved in any other research trials.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
The Scoliosis Research Society - 22r (SRS-22r) | baseline, 6 months and 12 months
  Patient reported outcome measure, measuring change in quality of life scores over 12 months.
  There are 22 questions within this outcome measure, which cover a variety of domains including:
  pain, body image, activity levels, function, mental health and social interaction.
  There are 5 scale points within each answer, but these 5 options are different each question.
  An example would be:
  1. Which one of the following best describes the amount of pain you have experienced during the past 6 months?
  None, Mild, Moderate, Moderate to severe, Severe.
  The most positive answer would be scored as 5 whilst the most negative answer would be scored 1. This process is consistent throughout the 22 questions and the scores of all 22 questions are added together for an overall score. A higher score suggests a higher quality of life.
  All of the questions in this outcome measure are designed to be scoliosis specific.

SECONDARY OUTCOMES:
The Short Form 36 point questionnaire (SF-36) | baseline, 6 months and 12 months
  A patient reported outcome measure, designed to measure quality of life using several sub-categories.
  This outcome measure is a questionnaire of 36 questions in total. It looks at:
  General health, limitations of activities, physical restrictions, social activities and pain.
  Each section has a different number of questions within it. Some questions have 5 scale points, some 3 and some 2.
  Within each question, the more negative answers are given the lower scoring and the more positive answers are given a higher scoring (which varies between 1-2, 1-3 and 1-5 depending on the question).
  The scores are then all added together for a total score. A higher total score indicates a higher quality of life and a lower total score indicates a lower quality of life.
The pain self-efficacy scale (PSES) | baseline, 6 months and 12 months
  A patient reported outcome measure which measures confidence in relation to performing certain tasks if in pain.
  There are two separate scales - one for the patient and one for the parent/guardian to complete. Both scales consist of 7 questions regarding levels of confidence performing certain functional tasks whilst being in pain. The scale ranges on each question are as follows:
  1 = Very Sure, 2 = Pretty Sure, 3 = In the middle, 4 = pretty unsure, 5 = very unsure.
  1 (very sure) is considered the best outcome. The scores from each question would be added together and therefore a lower overall sore is considered a better outcome.
The Global Rating of Change Scale (GRCS) | 6 months and 12 months post-operatively.
  A brief patient reported outcome measure, measuring level of overall change - in this case, whether the patient feels better or worse compared to just before their operation, and how much better or worse they feel.
  The scale ranges are:
  Better, No Change, or Worse.
  Within 'Better' there are then 5 sub-scale ranges which are:
  Slightly better, Somewhat better, Moderately better, Much better, very much better.
  Within 'Worse' there are 5 sub-scale ranges which are:
  Very much worse, much worse, moderately worse, somewhat worse, slightly worse.
  The scale is not numerical and will therefore give a guide for general/overall change since surgery rather than giving numerical data that is added up or averaged.

CONTACTS AND LOCATIONS:
Overall Officials: Jodie Walters, Principal Investigator — Physiotherapist
Locations (1):
- The Royal Orthopaedic Hospital NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adobor RD, Rimeslatten S, Keller A, Brox JI. Repeatability, reliability, and concurrent validity of the scoliosis research society-22 questionnaire and EuroQol in patients with adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2010 Jan 15;35(2):206-9. doi: 10.1097/BRS.0b013e3181b43bdf. PMID 20081517
- [Background] Bursch B, Tsao JC, Meldrum M, Zeltzer LK. Preliminary validation of a self-efficacy scale for child functioning despite chronic pain (child and parent versions). Pain. 2006 Nov;125(1-2):35-42. doi: 10.1016/j.pain.2006.04.026. Epub 2006 Jun 5. PMID 16740360
- [Background] Chan CYW, Aziz I, Chai FW, Kwan MK. A Silver Medal Winner at the 13th World Wu Shu Championship 2015 17 Months After Selective Thoracic Fusion for Adolescent Idiopathic Scoliosis: A Case Report. Spine (Phila Pa 1976). 2017 Feb 15;42(4):E248-E252. doi: 10.1097/BRS.0000000000001748. PMID 28207671
- [Background] Danielsson AJ, Wiklund I, Pehrsson K, Nachemson AL. Health-related quality of life in patients with adolescent idiopathic scoliosis: a matched follow-up at least 20 years after treatment with brace or surgery. Eur Spine J. 2001 Aug;10(4):278-88. doi: 10.1007/s005860100309. PMID 11563612
- [Background] Fabricant PD, Admoni S, Green DW, Ipp LS, Widmann RF. Return to athletic activity after posterior spinal fusion for adolescent idiopathic scoliosis: analysis of independent predictors. J Pediatr Orthop. 2012 Apr-May;32(3):259-65. doi: 10.1097/BPO.0b013e31824b285f. PMID 22411331
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Kim YJ, Lenke LG, Kim J, Bridwell KH, Cho SK, Cheh G, Sides B. Comparative analysis of pedicle screw versus hybrid instrumentation in posterior spinal fusion of adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2006 Feb 1;31(3):291-8. doi: 10.1097/01.brs.0000197865.20803.d4. PMID 16449901
- [Background] Lehman RA Jr, Kang DG, Lenke LG, Sucato DJ, Bevevino AJ; Spinal Deformity Study Group. Return to sports after surgery to correct adolescent idiopathic scoliosis: a survey of the Spinal Deformity Study Group. Spine J. 2015 May 1;15(5):951-8. doi: 10.1016/j.spinee.2013.06.035. Epub 2013 Oct 5. PMID 24099682
- [Background] Snowdon M, Peiris CL. Physiotherapy Commenced Within the First Four Weeks Post-Spinal Surgery Is Safe and Effective: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2016 Feb;97(2):292-301. doi: 10.1016/j.apmr.2015.09.003. Epub 2015 Sep 25. PMID 26409101
- [Background] Tones M, Moss N, Polly DW Jr. A review of quality of life and psychosocial issues in scoliosis. Spine (Phila Pa 1976). 2006 Dec 15;31(26):3027-38. doi: 10.1097/01.brs.0000249555.87601.fc. PMID 17173000
- [Background] Tsutsui S, Pawelek J, Bastrom T, Lenke L, Lowe T, Betz R, Clements D, Newton PO. Dissecting the effects of spinal fusion and deformity magnitude on quality of life in patients with adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2009 Aug 15;34(18):E653-8. doi: 10.1097/BRS.0b013e3181b2008f. PMID 19680091
- [Background] Yu CH, Chen PQ, Ma SC, Pan CH. Segmental correction of adolescent idiopathic scoliosis by all-screw fixation method in adolescents and young adults. minimum 5 years follow-up with SF-36 questionnaire. Scoliosis. 2012 Feb 19;7:5. doi: 10.1186/1748-7161-7-5. PMID 22340624